CLINICAL TRIAL: NCT05523648
Title: Clinical Effects of Ganshuang Combined TDF to Treat CHB and NAFLD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan Leshan Traditional Chinese Medicine Hospital (Other)
Responsible Party: Principal Investigator, Qin Yang, Deputy chief physician, Sichuan Leshan Traditional Chinese Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Qin1651
Record Dates: First submitted 2022-08-24; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis B; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Experimental): The control group was treated with silibinin meglumine tablets and tenofovir
  Interventions: Drug: Chronic Hepatitis B
- The treatment group (Active Comparator): The treatment group was treated with Ganshuang granules combined with silibinin meglumine tablets and tenofovir
  Interventions: Drug: Chronic Hepatitis B

INTERVENTIONS:
Drug: Chronic Hepatitis B — 92 patients included in the study were randomly divided into 2 groups, 42 patients in the control group and 50 patients in the treatment group. Both groups of patients received conventional basic treatment such as liver protection. Moreover, in both groups, patients were instructed to change their dietary structure to control low-fat and low-sugar, and were instructed to perform appropriate aerobic exercise.
  Other Names: Nonalcoholic Fatty Liver Disease

SUMMARY:
The changes in liver function, body mass index, controlled attenuation parameters, liver stiffness and HBV-DNA at different time points in each group before and after treatment were counted to explore the clinical efficacy of Ganshuang granules combined with tenofovir in the treatment of CHB complicated with NAFLD.

DETAILED DESCRIPTION:
92 patients included in the study were randomly divided into 2 groups, 42 patients in the control group and 50 patients in the treatment group. Both groups of patients received conventional basic treatment such as liver protection. Moreover, in both groups, patients were instructed to change their dietary structure to control low-fat and low-sugar, and were instructed to perform appropriate aerobic exercise.

The control group was treated with silymarin glucosamine tablets (Jiangsu Zhongxing Pharmaceutical Co., Ltd.; National medicine permission number: H32026233; Production batch: 200304) and tenofovir (QILU Pharmaceutical Co., Ltd.; National medicine permission number: H20173185; Production batch: 1L0694DF6). The use of silymarin glucosamine tablets was 0.2g/d, 3 times/d for 24 weeks; the use of tenofovir was 300mg/d, 1 time/d for 24 weeks.

The treatment group was treated with Ganshuang granules (Baoding Tianhao Pharmaceutical Co., Ltd.; National medicine permission number: Z20027671; Production batch: 200326 ) combined with silibinin meglumine tablets and tenofovir. Libribin meglumine tablets and tenofovir were used in the same way as in the control group, and Ganshuang granules were used 3 g/time, 3 times/d, and the course of treatment was 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

Chronic hepatitis B patients not treated with antiviral drugs； Fatty liver was diagnosed by B-ultrasound and imaging； No history of excessive drinking； Good drug compliance and regular medication； Exclusion Criteria： Non chronic hepatitis B patients； Taking other drugs； liver failure, liver cancer and other diseases； patients who refused to sign informed consent；

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
ALT, AST and GGT | 12 and 24 weeks
  Alt, AST and GGT were used to evaluate the improvement of liver function before and after treatment
HBV-DNA serum load < 500 IU/ml | 12 and 24 weeks
  To verify the effect of the drug on the clearance of hepatitis B virus, the number of patients with HBV-DNA serum load < 500 IU/ml before and after treatment was counted in this study
liver stiffness | 12 and 24 weeks
  In our study, liver sclerosis index was detected using LSM to compare the improvement of liver stiffness before and after treatment in the two groups
fat attenuation | 12 and 24 weeks
  The LSM was used to detect and compare fat attenuation parameters in this study

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yang, MM, Study Chair — Sichuan Leshan Traditional Chinese Medicine Hospital
Locations (1):
- Sichuan Leshan traditional Chinese medicine hospital, Leshan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su C, Yang Q. Clinical study of ganshuang granule combined with tenofovir in the treatment of chronic hepatitis B complicated with nonalcoholic fatty liver disease. Front Pharmacol. 2022 Dec 14;13:1032789. doi: 10.3389/fphar.2022.1032789. eCollection 2022. PMID 36588741